CLINICAL TRIAL: NCT03247439
Title: A Prospective Study to Evaluate the Safety and Effectiveness of the Cartiva® Synthetic Cartilage Implant for CMC in the Treatment of First Carpometacarpal Joint Osteoarthritis as Compared to a Ligament Reconstruction Tendon Interposition (LRTI) Comparator
Brief Title: Safety and Effectiveness of Cartiva Implant in the Treatment of First CMC Joint Osteoarthritis Compared to LRTI (GRIP 2)
Acronym: GRIP 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC-0290
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis
Keywords: CMC Joint; Osteoarthritis; Cartilage Replacement; First CMC Joint Osteoarthritis; Damaged Articular Surface; LRTI; Ligament Reconstruction Tendon Interposition
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cartiva (Experimental): Synthetic Cartilage Implant
  Interventions: Device: Cartiva

INTERVENTIONS:
Device: Cartiva — Synthetic Cartilage Implant

SUMMARY:
This study will evaluate whether Cartiva is an effective treatment for individuals with osteoarthritis of the first CMC joint in the hand compared to LRTI.

DETAILED DESCRIPTION:
This is a prospective, multicenter study with one treatment arm. Comparisons will be made to a performance target defined by subtracting a non-inferiority margin of 0.05 from an expected standard of care success rate of 0.55. The active treatment arm will receive a Cartiva® SCI for CMC.

A total of 74 subjects will be enrolled into the pivotal study.

Follow up visits will occur at the following time points after the surgical procedure: 2 week, 6 week, 3 month, 6 month, 1 year, 2 year, 3 year, 4 year and 5 year.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 22 years of age
* Refractory to conservative non-operative standard of care treatment for first CMC OA lasting for at least 6 months that requires surgical intervention
* Eaton classification stage II or III OA of the first CMC joint based on X-rays taken within 6 months of the Operative date and evidence of first CMC joint OA based on subjective review of associated clinical symptoms
* Preoperative VAS Pain score of ≥ 40 in the treated hand
* Preoperative 11 question QuickDASH score of ≥ 20
* Presence of good bone stock - i.e., no need for bone graft
* Capable of completing self-administered questionnaires
* Be willing and able to return for all study-related follow up procedures
* Have been informed of the nature of the study, agreeing to its requirements, and have signed the informed consent approved by the IRB/REB/Ethics Committee

Exclusion Criteria:

* Active systemic infection
* Active infection at the site of surgery
* Previous CMC implant, trapeziectomy, or LRTI to the affected joint to be treated
* Inflammatory arthropathy and/or diagnosis of grout
* History of or current diagnosis of rheumatoid arthritis
* Any significant bone loss, avascular necrosis, or cyst > 8mm of the supporting bone structure
* Eaton classification stage IV advanced OA of the first CMC joint based on X-rays taken within 6 months of the Operative date
* Physical conditions that would tend to eliminate adequate implant support (e.g., inadequate cortical bone stock of at least 2mm circumferentially insufficient quality or quantity of bone resulting from cancer, congenital dislocation, or osteoporosis), systemic and metabolic disorders leading to progressive deterioration of bone (e.g., cortisone therapies or immunosuppressive therapies), and/or tumors and/or cysts of the supporting bone structures
* OA of the scaphotrapeziotrapezoidal (STT) joint based on radiographic assessment in the hand to be treated
* Any disease, including uncontrolled diabetes mellitus, which is clinically known to impact wound healing ability
* Known or suspected allergic reaction to polyvinyl alcohol
* Patient is on chronic anticoagulation due to a bleeding disorder or has taken anticoagulants within 3 days prior to surgery
* Diagnosed with cancer in the last two years and received treatment with chemotherapy or received radiation to the upper extremity to be treated with Cartiva
* Any medical condition that makes the subject unsuitable for inclusion in the study, including, but not limited to, patients with a diagnosis of concomitant injury that may interfere with healing; patients with clinically significant renal, hepatic, cardiac, endocrine, hematologic, autoimmune or any systemic disease or systemic infection which may make interpretation of the results difficult; patients who have undergone systemic administration within 30 days prior to implantation of any type of corticosteroid in the thumb, antineoplastic, immunostimulating or immunosuppressive agents
* Have participated in any other investigational or invasive clinical trial within the last three months, and will not participate in any other investigational or invasive clinical trial during this study
* Co-morbidity that reduces life expectancy to less than 12 months
* If female, be pregnant, planning to become pregnant during the course of the study, breast-feeding, or if childbearing age, is not using contraception
* Current or recent history of substance abuse (e.g., recreational drugs, narcotics, or alcohol) requiring intervention
* Is a prisoner or ward of the state
* Is unable to meet the treatment and follow up protocol requirements
* Is being compensated under workers' compensation or are currently involved in litigation that is related to the musculoskeletal system

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Pain measured by the Visual Analog Scale (VAS) scale | 1 year
  Success criteria: ≥ 30% VAS decrease at 12 months. Visual Analog Scale (VAS) Pain score will be obtained from the subject for pain in the treated hand by completing a CRF, which has a 100 mm horizontal line on it, with the left end indicating that the subject has no pain and the right end of the line indicating a lot of pain. The subject will be instructed to place a mark on the horizontal line to rate the average pain in the treated thumb joint over the past week. The designated site staff will use a metric ruler to measure the markings made by the subject on the VAS to determine the VAS score.
Function measured by QuickDASH | 1 year
  Success criteria: ≥ 15.9 point decrease at 12 months. QuickDASH functional score will be obtained from the subject. The QuickDASH, the shortened version of the DASH (Disabilities of the Arm, Shoulder, and Hand) Outcomes Measures, is a region-specific, self-reported questionnaire that uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. Subjects are asked to circle the appropriate response to each question based on their condition in the past week.
Radiographic Findings | 1 year
  Success criteria: Freedom from radiographic failures post-surgery through 12 months. Radiographic failures are defined as device dislocation, device fragmentation and/or development of avascular necrosis.
Key Subsequent Secondary Surgical Interventions (SSSIs) | 1 year
  Success criteria: Freedom from Subsequent Secondary Surgical Interventions (SSSIs) through 12 months. SSSIs are defined as revisions, removals, reoperations, and/or supplemental fixations.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wolfe, MD, Principal Investigator — Hospital for Special Surgery, New York; Christopher Bainbridge, MB ChB, FRCSEd, CCST, Principal Investigator — Royal Derby Hospital
Locations (9):
- United States (5):
  - University of California, San Diego, San Diego, California
  - Georgia Hand, Shoulder & Elbow, Atlanta, Georgia
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Hospital for Specialty Surgery, New York, New York
  - University of Rochester, Rochester, New York
- United Kingdom (4):
  - Royal Derby Hospital, Derby, Derbyshire
  - Dorset County Hospital, Dorchester, Dorset
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - South Tees Hospitals, Middlesbrough, North Yorkshire

IPD SHARING:
Plan to Share IPD: No